CLINICAL TRIAL: NCT06925438
Title: Comparison Between Computer Guided and Free Hand Placement of Zygomatic Implants (Clinical and Radiographic Evaluation)
Brief Title: "Computer-Guided vs Freehand Zygomatic Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdelfattah Moawad Abdelfattah, Assistant Lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZygomaticRCT880/62
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dental Implants; Maxillary Diseases
Keywords: "Zygomatic implants"; "Atrophic maxilla rehabilitation"; "Guided implant surgery"; "Free-hand dental implantation"; "3D-printed surgical guides"
MeSH Terms: conditions — Maxillary Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: "The participants, care providers, and outcomes assessors were blinded to the method of implant placement (computer-guided or freehand) to minimize bias."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computer-Guided Zygomatic Implants (Active Comparator): Zygomatic implants placed using 3D-printed bone-supported surgical guides created from preoperative CT scans.
  Interventions: Procedure: Computer-guided zygomatic implant system
- Free-Hand Zygomatic Implants (Placebo Comparator): Zygomatic implants placed using anatomical landmarks (ZAGA classification) without surgical guides.
  Interventions: Procedure: free-hand zygomatic implant placement

INTERVENTIONS:
Procedure: Computer-guided zygomatic implant system — Preoperative digital planning (DICOM data) to fabricate guides with metal sleeves for drill alignment
  Arms: Computer-Guided Zygomatic Implants
Procedure: free-hand zygomatic implant placement — Standard placement using sequential drills (2.8-3.6mm) under saline irrigation
  Arms: Free-Hand Zygomatic Implants

SUMMARY:
This randomized trial compares computer-guided versus free-hand zygomatic implant placement in patients with atrophic maxillae or maxillary defects. Participants receive either 3D-navigated implants (using stereolithographic guides) or conventional free-hand placement. Primary outcomes measure accuracy through apical angular deviation (°), apical/coronal linear deviations (mm) relative to MSP/FHP/CP planes (CT-based), while secondary outcomes assess implant stability (ISQ) and complications (sinusitis/infection) over 6 months. The study evaluates whether guided surgery improves precision in complex maxillary rehabilitation.

DETAILED DESCRIPTION:
"This study was retrospectively registered due to initial lack of awareness of prospective registration requirements. All procedures followed ethical guidelines (Approval #880/62), and results are reported transparently."

Study Design

A single-center, randomized controlled trial conducted at Al-Azhar University, comparing computer-guided versus free-hand zygomatic implant placement. Participants are allocated 1:1 to:

Group A (Free-hand): Implants placed using ZAGA classification with conventional surgical techniques.

Group B (Guided): Implants placed via 3D-printed bone-supported surgical templates (DICOM-based planning).

Interventions

Both Groups:

Pre-op: CT scans for zygomatic bone assessment.

Anesthesia: General anesthesia with local infiltration for hemostasis.

Surgical Protocol: Full-thickness flap, implant placement , two-stage healing.

Group B-Specific Steps:

Digital implant path planning (entrance/exit points).

Stereolithographic guide fabrication with metal sleeves.

Guide fixation with monocortical screws during surgery.

Rationale Zygomatic implants require high precision due to anatomical complexity. While free-hand placement depends on surgeon skill, computer guidance may reduce errors. This trial evaluates whether guided surgery improves accuracy (angular deviation) and reduces complications (sinusitis, infection).

Methodological Rigor Randomization: Block randomization via SPSS.

Blinding: Radiographic assessors blinded to group allocation.

Sample Size: 16 implants (8/group), powered to detect 3.73° mean angular deviation difference (α=0.05, β=0.10; based on Grecchi et al. 2022).

Ethical Compliance Approved by Al-Azhar University (Ref: 880/62).

Consent forms documented risks/benefits (e.g., sinus perforation, infection).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years
* Atrophic maxillary ridge (Cawood & Howell Class IV-VI)
* Maxillary defects due to trauma, tumor resection, or congenital conditions

Exclusion Criteria:

* Acute maxillary sinusitis
* Uncontrolled systemic diseases affecting osseointegration
* Pathological lesions in maxilla/zygoma
* Heavy smoking (>20 cigarettes/day)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Angular deviation of zygomatic implants | Measured immediately post-operatively (Day 0)
  Difference in degrees between planned (virtual) and actual post-operative implant position, measured at the apical point using superimposed CT scans
Apical linear deviation of zygomatic implants | Measured immediately post-operatively (Day 0)
  Difference in millimeters between planned (virtual) and actual post-operative implant position at the apical point, measured using superimposed CT scans along three planes midsagittal plane (MSP) - Frankfort horizontal plane (FHP) - coronal plane (CP)
Coronal linear deviation of zygomatic implants | Measured immediately post-operatively (Day 0)
  Difference in millimeters between planned and actual implant position at the coronal point (implant neck), measured using superimposed CT scans along three planes midsagittal plane (MSP) - Frankfort horizontal plane (FHP) - coronal plane (CP)

SECONDARY OUTCOMES:
Implant stability quotient (ISQ) | Immediately post-op and at 6 months
  Primary and secondary stability measured using Osstell Mentor device at implant placement and 6-month follow-up"
Postoperative complication rates | Assessed at 1 week, 1 month, 3 months, and 6 months post-op
  Incidence of sinusitis, infection, soft tissue dehiscence, and oroantral communication assessed clinically

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa El-Din Abd Raboo, phd, Study Director — Al-Azhar University, faculty of dentistry ,Oral & Maxillofacial Surgery Dept; Mohamed Abdel Akhar, PhD, Study Director — Al-Azhar University, faculty of dentistry, Oral & Maxillofacial Surgery Dept; Abdelfattah Moawad, BDS, MSc, Principal Investigator — Al-Azhar University, faculty of dentistry, Oral & Maxillofacial Surgery Dept
Locations (2):
- Egypt (2):
  - Faculty of Dental Medicine - Boys, Al-Azhar University, Cairo, Cairo Governorate
  - Oral and Maxillofacial Surgery Department, Faculty of Dental Medicine - Boys, Al-Azhar University, Cairo, Cairo Governorate

IPD SHARING:
Plan to Share IPD: No
Data is available with corresponding offer on reasonable request